CLINICAL TRIAL: NCT04457076
Title: A Phase 3, Prospective, Multi-Center, Single-Arm, Open-Label Study to Evaluate LevoCept™, a Long-Acting Reversible Intrauterine System for Contraceptive Efficacy, Safety, and Tolerability
Brief Title: Evaluation of the Efficacy, Safety, and Tolerability of LevoCept
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sebela Women's Health Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: Sebela Pharmaceuticals Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMDOC-0062
Record Dates: First submitted 2020-06-11; First posted 2020-07-07 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Contraception; Women at Risk for Pregnancy
Keywords: Contraception; IUD

STUDY DESIGN:
Intervention Model Description: LevoCept Intrauterine Device (IUD)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LevoCept (Experimental): LevoCept™ Intrauterine Contraceptive
  Interventions: Drug: LevoCept

INTERVENTIONS:
Drug: LevoCept — Levonorgestrel-Releasing Intrauterine System

SUMMARY:
To assess the contraceptive efficacy (prevention of pregnancy) of LevoCept

DETAILED DESCRIPTION:
Study Design:

Prospective, multi-center, single-arm, open-label, Phase 3 clinical study to 3 years with extension up to 5 years

Number of Subjects:

Approximately 1,525 subjects will be enrolled into the study

Study Population:

Post-menarcheal, pre-menopausal women up to age 45 years, who are at risk for pregnancy and who desire a long-term intrauterine contraceptive for birth control will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menarcheal, pre-menopausal females up to 45 years of age at the time of informed consent/assent and in good general health;
2. History of regular menstrual cycles defined as occurring every 21-35 days when not using hormones or prior to recent pregnancy or spontaneous or induced abortion;
3. Sexually active with a male partner who has not had a vasectomy nor other known fertility problems;
4. Reasonably expect to have coitus at least once monthly during the study period;
5. In a mutually monogamous relationship of at least 3 months duration at time of consent;
6. Seeking to avoid pregnancy for the duration of the study;
7. Willing to use the study drug as the sole form of contraception;
8. Willing to accept a risk of pregnancy;
9. Subjects must be in compliance with cervical cancer screening guidelines per the American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines without evidence of disease. Subjects who are age 21 to 24 y/o, at time of informed consent, must have a normal Papanicolaou test (Pap), atypical squamous cells of undetermined significance (ASC-US), or low-grade squamous intraepithelial lesion (LSIL). Subjects who are 25 or older at the time of informed consent must have a normal Pap test or an ASC-US result with a negative high-risk human papilloma virus (HPV) test result within the appropriate screen timeframe per ASCCP guidelines, and prior to the study IUD insertion. Alternatively, the subject must have had a colposcopy performed within the appropriate screen timeframe, and prior to the study IUD insertion that showed no evidence of dysplasia requiring treatment per ASCCP guidelines, or treatment was performed and follow-up at least 6 months after the treatment showed no evidence of disease by clinical evaluation;
10. Able and willing to comply with all study tests, procedures, assessment tools (including e-diary) and follow-up;
11. Able and willing to provide and document informed consent and Authorization for Release of Protected Health Information (PHI). Unemancipated subjects under 18 years old must provide assent and have written parental/legal guardian consent documented on the consent form consistent with local legal requirements;
12. Plan to reside within a reasonable travel distance of a research site for the duration of the study.
13. Subject agrees not to intentionally self-remove LevoCept

Exclusion Criteria:

1. Known or suspected pregnancy; or at risk for pregnancy from unprotected intercourse earlier in current cycle;
2. Has had any procedure for or causing sterility (e.g. tubal ligation procedure);
3. Subject who anticipates separation from her partner for more than a 6-month period during use of LevoCept;
4. A previously inserted IUD/IUS that has not been removed by the time the study IUS is placed;
5. History of previous IUD/IUS complications, such as perforation, expulsion, or pregnancy with IUD/IUS in place;
6. Pain with current IUD/IUS;
7. Injection of hormonal contraceptive (e.g., Depo-Provera) within the last 10 months and has not had 2 normal menstrual cycles since the last injection;
8. Subject is <4 weeks post-pregnancy (postpartum, spontaneous or induced abortion)
9. Planned use of any non-contraceptive estrogen, progesterone or testosterone any time during the 60 months of study participation;
10. Exclusively breastfeeding before return of menses; lactating women will be excluded unless they have had 2 normal menstrual periods prior to enrollment;
11. Unexplained abnormal uterine bleeding (suspicious for a serious condition), including bleeding 4 weeks post-septic abortion or puerperal sepsis;
12. Severely heavy or painful menstrual bleeding;
13. Suspected or known cervical, uterine or ovarian cancer, or unresolved clinically significant abnormal Pap test requiring evaluation or treatment;
14. Any history of gestational trophoblastic disease with or without detectable elevated ß-human chorionic gonadotropin (ß-hCG) levels, or related malignant disease;
15. Any congenital or acquired uterine anomaly that may complicate study drug placement, such as:

    * Submucosal uterine leiomyoma
    * Asherman's syndromes
    * Pedunculated polyps
    * Bicornuate uterus
    * Didelphus or uterine septa
16. Any distortions of the uterine cavity (e.g. fibroids), that, in the opinion of the investigator, are likely to cause issues during insertion, retention or removal of the IUS;
17. Known anatomical abnormalities of the cervix such as severe cervical stenosis, prior trachelectomy or extensive conization that, in the opinion of the investigator would prevent cervical dilation and study drug placement;
18. Untreated or unresolved acute cervicitis or vaginitis;
19. Known or suspected breast cancer or other progestin-sensitive cancer now or in the past;
20. Known acute liver disease or liver tumor;
21. Subjects who have an established immunodeficiency;
22. Known or suspected human immunodeficiency virus (HIV) infection or clinical AIDS;
23. At high risk for sexually transmitted infections (e.g. multiple sexual partners);
24. Known intolerance or allergy to any components of LevoCept, including intolerance or allergy to levonorgestrel, nickel, titanium, or silicone;
25. Currently participating or planning future participation in a research study of an investigational drug or device during the course of this investigational study. Subject must have waited at least 30 days from exiting their last study prior to informed consent in this study;
26. Subject has previously been enrolled in a VeraCept or LevoCept study (including the current study);
27. Known or suspected alcohol or drug abuse within 12 months prior to the screening visit;
28. Any general health, mental health or behavioral condition that, in the opinion of the investigator, could represent an increased risk for the subject or would render the subject less likely to provide the needed study information;
29. Study staff or a member of the immediate family of study staff.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1525 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Contraceptive efficacy through 3 years of use as calculated by the Pearl Index | through 3 years of use

SECONDARY OUTCOMES:
Contraceptive efficacy at Years 4 and 5 as calculated by the Pearl Index | Years 4 and 5 and cumulatively through Years 4 and 5
Pregnancy percentage | Years 1 through 5
Ease of LevoCept placement | Day 1 / LevoCept placement
  Ease of LevoCept placement will be summarized for the Safety population as reported by the investigator (Very easy, Easy, Neither Easy nor Hard, Hard, Very Hard).
LevoCept Placement success | Day 1 / LevoCept placement
  The number of subjects with either a successful or unsuccessful placement will be summarized
Incidence of AEs and SAEs | 5 years
Bleeding and spotting patterns | Through year 1
Insertion pain assessed immediately after insertion | Day 1, immediately after insertion
  Summarized for subjects with and without prior prophylactic pain medication as measured by an 11-Point Numeric Pain Rating Scale. The scale being 0 - 10 with 0 being no pain and 10 being the worse pain
Cumulative LevoCept continuation rates | Years 1 through 5
  Continuation rates at Years 1, 2, 3, 4 and 5, Reasons for discontinuation will be summarized.
Cumulative LevoCept expulsion rates | Years 1 through 5
Return to Fertility. Only for subjects requesting LevoCept removal to become pregnant. | Subjects will be followed for either 1 year, until they decide to no longer try to conceive or they become pregnant, whichever comes first.
Release rate of LNG from the IUS and resulting pharmacokinetics of LNG (PK substudy) | Years 1 through 5

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Essential Access Health-Berkeley, Berkeley, California
  - Essential Access Health-Los Angeles, Los Angeles, California
  - University of California Davis Health System Department of Obstetrics and Gynecology, Sacramento, California
  - WR-Medical Center for Clinical Research, San Diego, California
  - Women's Health Care Research, San Diego, California
  - Stanford University, Medical Center, Obstetrics and Gynecolocy, Stanford, California
  - University Of Colorado Department of Obstetrics & Gyncology, Aurora, Colorado
  - Emory University School of Medicine Gynecology/Obstetrics, Atlanta, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - IU Health University Hospital, Indianapolis, Indiana
  - Planned Parenthood North Central States, Minneapolis, Minnesota
  - Planned Parenthood of the St. Louis Region and Southwest Missouri, Manchester, Missouri
  - Rex Garn Mabey Jr., MD, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati/Reproductive Medicine Research, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - The Ohio State University Ob/Gyn Research Office, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Center for Family Planning Research, Pittsburgh, Pennsylvania
  - Advances In Health, Houston, Texas
  - University of Utah Healthcare Health Sciences Center, Salt Lake City, Utah
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Eastern Virginia Medical, Norfolk, Virginia
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No